CLINICAL TRIAL: NCT06889298
Title: Safety and Efficacy of the BTL-699 Device for Temporary Reduction of Food Cravings
Brief Title: EXOMIND (BTL-699) for the Reduction of Food Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-699_CTCZ100
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-03

CONDITIONS: Food Cravings
Keywords: rTMS; food cravings; weight reduction; ExoTMS; EXOMIND
MeSH Terms: conditions — Weight Loss | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with BTL-699 (Experimental): Transcranial magnetic stimulation treatments with the BTL-699 device
  Interventions: Device: Treatment with BTL-699

INTERVENTIONS:
Device: Treatment with BTL-699 — Four to six transcranial magnetic stimulation treatments with the BTL-699 device will be delivered over the left dorsolateral prefrontal cortex, spaced 2 to 3 days apart. The intensity will be adjusted according to the subject's feedback, up to 100% of the individual's motor threshold.
  Other Names: EXOMIND (BTL-995) with ExoTMS

SUMMARY:
The goal of this clinical trial is to evaluate if the treatment with BTL-699 device is able to temporarily reduce food cravings in adults above the age of 22 years. The main question it aims to answer is:

Does the treatment with BTL-699 device provide a temporary reduction of food cravings?

Participants will be asked to:

* Undergo 4 to 6 treatments
* Undergo weight measurements
* Complete the Food Cravings Questionnaire-Trait
* Complete the Therapy Comfort Questionnaire
* Complete the Satisfaction Questionnaire

DETAILED DESCRIPTION:
This study uses a single-center, single-arm, open-label, interventional design.

Subjects reporting at least 3 to 5 weekly instances of food cravings will be enrolled. All enrolled participants will receive 4 to 6 treatments with the BTL-699 device, administered 2 to 3 days apart. The required number of treatments for each participant will be determined on a case-by-case basis by the Principal Investigator, with a minimum of four sessions.

Therapy parameters will be adjusted based on patient feedback and comfort, up to 100% of the individual's motor threshold.

Examination for possible adverse effects will be assessed at each visit.

The Food Cravings Questionnaire-Trait will be administered before the first treatment, after the last treatment, and at the two follow-up visits-2 weeks and 1 month after the final session.

The Therapy Comfort Questionnaire will be administered after the last treatment, while the Satisfaction Questionnaire will be given after the last treatment and at both follow-up visits.

The total expected duration of subject participation, from the baseline visit to study completion, is approximately three months.

ELIGIBILITY:
Inclusion Criteria:

* At least 3-5 self-reported episodes of food craving periods per week
* Age > 22 years
* Ability to determine the motor threshold of the participant. The participant's motor threshold could be established as the minimum stimulus required to induce contraction of the right thumb at least five out of 10 times
* Subjects willing and able to abstain from partaking in any other weight management treatments other than the study procedure during study participation
* Willingness to comply with study instructions and to return to the clinic for the required visits

Exclusion Criteria:

* Cochlear implants
* Intake disorders such as bulimia, anorexia
* Borderline personality disorder
* Other metal implants close to the application area (1 meter at least)
* Personal history of epilepsy
* Personal history of syncope
* Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without a history of seizure, and without anticonvulsant medication
* Sleep deprivation
* Alcoholism
* Presence of a substance abuse or dependence (alcohol, caffeine, drugs) conditions associated with altered seizure risk
* Intake of one or a combination of the following drugs forms a strong potential hazard for the application of rTMS due to their significant seizure threshold lowering potential: imipramine, amitriptyline, doxepine, nortriptyline, maprotiline, chlorpromazine, clozapine, foscarnet, ganciclovir, ritonavir, amphetamines, cocaine, (MDMA, ecstasy), phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), alcohol, theophylline
* Intake of seizure threshold lowering drugs such as: mianserin, fluoxetine, fluvoxamine, paroxetine, sertraline, citalopram, reboxetine, venlafaxine, duloxetine, bupropion, mirtazapine, fluphenazine, pimozide, haloperidol, olanzapine, quetiapine, aripiprazole, ziprasidone, risperidone, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, BCNU, lithium, anticholinergics, antihistamines, sympathomimetics
* Withdrawal from one of the following drugs could form a relative hazard for the application of rTMS due to the resulting significant seizure threshold lowering potential: alcohol, barbiturates, benzodiazepines, meprobamate, chloralhydrate
* Systemic infection, fever
* Patients with a broad range of neuropsychiatric diseases are at elevated risk for seizures. - Essentially all neurologic conditions with structural cerebral damage (e.g. stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers) are associated with an elevated risk for seizures
* Major depression (elevated seizure risk)
* Hyponatremia, hypocalcemia, hypomagnesemia, hypoglycemia, hyperglycemia, renal failure/uremia, liver failure
* Raised blood concentrations of pro-convulsant medications due to reduced clearance (e.g. secondary to initiation of antibiotics for treatment of infections)
* Immunosuppressive therapy with cyclosporine, tacrolimus and other agents that can cause the posterior reversible leukoencephalopathy syndrome
* Dialysis
* Bipolar Disorder
* Pregnancy or lactation, absence of medically approved contraceptive methods in females of childbearing potential
* Urine drug screen positive for amphetamines, barbiturates, cannabinoids, cocaine metabolites, opiates and phencyclidine
* Implanted infusion pumps
* Intracardiac devices (pacemakers, heart valves, etc.)
* Contradictions for the testing used in the trial, for example, the motor threshold cannot be found or quantified

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in Food Cravings | 15 months
  The change in the score obtained from the Food Cravings Questionnaire-Trait will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, at the 2-week and 1-month follow-up visits. The score ranges from 39 to 234 and higher scores indicate more frequent and intense food cravings in general. An improvement is defined as a decrease in score.

SECONDARY OUTCOMES:
Assessment of Therapy Comfort | 15 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the last treatment. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree") and the 10-point Numeric Analog Scale for pain (0 = no pain, 10 = worst possible pain"). A higher score for the statement "I found the treatment comfortable", and lower score on the Numeric Analog Scale for pain indicate higher therapy comfort.
Assessment of Satisfaction | 15 months
  Subject Satisfaction with treatment outcomes will be assessed using 5-point Likert Scale Satisfaction questionnaire. The questionnaire will be administered after the last treatment, at the 2-week and 1-month follow-up visits. Responses to questions about satisfaction with the treatment outcomes will range from "strongly agree" (5 points) to "strongly disagree" (1 point). A higher score for each statement indicate better outcomes.
Incidence of Treatment-related Adverse Events | 15 months
  Monitoring of adverse reactions and side effects will be performed for the evaluation of safety of the treatment with the BTL-699 device for the reduction of food cravings and to identify side effects and adverse events associated with the study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute for Mental Health, Klecany, Czechia